CLINICAL TRIAL: NCT03542968
Title: Imaging by 4 DFlow in Patients With Tetralogy of Fallot
Acronym: 4DFlowFallot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A01482-51
Record Dates: First submitted 2018-05-04; First posted 2018-06-01 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2019-06

CONDITIONS: Congenital Heart Disease
Keywords: Congenital heart disease; Tetralogy of Fallot; Imaging by 4D Flow,; Magnetic resonance imaging; Prevention of ventricular dysfunction
MeSH Terms: conditions — Heart Defects, Congenital; Tetralogy of Fallot | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4D magnetic resonance imaging (Experimental): MRI, 4D imaging, acquisition and analysis of 4D cardiac MRI images-A single, faster acquisition (8 to 15 minutes).
  Interventions: Procedure: magnetic resonance imaging
- 2D magnetic resonance imaging (Sham Comparator): MRI, 2D imaging, acquisition and analysis of 2D cardiac MRI
  Interventions: Procedure: magnetic resonance imaging

INTERVENTIONS:
Procedure: magnetic resonance imaging — Acquisition 4D Flow magnetic resonance Imaging-8 minutes

SUMMARY:
Conventionnal cadiac magnetic resonance (CMR) is the reference to assess changes in right heart flow and pulmonary artery hemodynamics in patients with repaired Tetralogy of Fallot.

4D Flow CMR Imaging is a new imaging modality able to assess all of these parameters faster (8 min vs 30 min) and more comfortably.

The aim of this study is to compare conventionnal CMR and 4D Flow CMR for the assessment of these parameters (ventricular volume, ventricular systolic function, and regurgitation of the pulmonary pathway).

DETAILED DESCRIPTION:
Congenital heart disease, or corrected heart disease requires regular, specialized follow-up throughout the life of these patients. Among the recommended examinations, cardiac MRI is the reference for functionnal ventricles assessment (volume/systolic function), particularly for the right ventricle.

Among these pathologies, the tetralogy of Fallot is indicative of the increasing importance of cardiac MRI. In this disease, strong parameters has been identifies for the follow to prevent right ventricle dysfunction and ventricular arrhythmias. They rely on right ventricle volumes and on the pulmonary artery regurgitation, both using cardiac MRI.

However, this imaging modality imposes constraints such as a long acquisition times (30 to 40 min) or the need to hold apneas, which may render the procedure uncomfortable, even more in the case of very young patients.

The idea of exploring a new imaging modality is therefore based on the willingness to offer a faster and more comfortable examination. 4D Flow MRI could enable conventionnal parameters, detection of both normal and abnormal right heart flow patterns, and may allow comprehensive analysis of post-surgically altered geometries and hemodynamics.

4D Flow MRI cardiac imaging is :

* A single and faster acquisition (8 to 15 minutes) that cardiac MRI.
* A free breathing acquisition Imaging modality.
* A quite-isotropic assessment.
* A technically simple exam (a single sequence requiring low competence).
* And offers unlimited post processing.

The investigators hypothesize that 4D MRI is non-inferior to 2D MRI in patients with corrected tetralogy of Fallot, for the evaluation of conventional cardiac evaluation parameters: ventricular volume, ventricular systolic function, and regurgitation of the pulmonary pathway.

The investigators hypothesize that 4D MRI is superior to 2D MRI in patients with corrected tetralogy of Fallot, as ti allows to identifying new predictors of ventricular dysfunction such as intravenous extracardiac turbulent / laminar flow character, preferential orientation, flow distribution and trans-tricuspid diastolic flow.

ELIGIBILITY:
Inclusion Criteria:

* - children from the age of 10 and above without any upper age limit;
* giving their informed consent for the study;
* with a corrected tetralogy of Fallot;
* sent for a follow-up imaging examination with endomyocardial fibrosis screening;

Exclusion Criteria:

* - pregnant woman;
* children <10 years old;
* All contraindications inherent to MRI: (claustrophobia, ferromagnetic intracorporeal foreign bodies)
* Contraindication to contrast media injection (Gadolinium)

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-10-12 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2020-04-11 (Estimated)

PRIMARY OUTCOMES:
Comparison of the pulmonary artery regurgitation using 2D MRI and 4D Flow MRI. | 20 min
  Assessment of the pulmonary artery regurgitation using 2D MRI and 4D Flow MRI : regurgitation volume (ml) and regurgitation fraction (%).

SECONDARY OUTCOMES:
Compare the evaluation of right ventricle volumes using 2D MRI and 4D Flow MRI. | 20 min
  Assessment of the end-diastolic and end-systolic right ventricle volumes using 2D MRI and 4D Flow MRI (ml).

CONTACTS AND LOCATIONS:
Overall Officials: Marc Antoine ISORNI, Doctor, Principal Investigator — Hôpital Marie Lannelongue
Locations (1):
- Hôpital Marie Lannelongue, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: No